CLINICAL TRIAL: NCT07144917
Title: Immunoparalysis After Pancreaticoduodenectomy : a Pilot Multicentric Prospective Study Based on mHLA-DR Expression
Brief Title: Immunoparalysis After Pancreaticoduodenectomy
Acronym: ImPaHLA
Status: Not yet recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_1056
Record Dates: First submitted 2025-08-20; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Ductal Adenocarcinoma (mPDAC); Pancreatic Head Tumour; Pancreatic Fistula
Keywords: Pancreaticoduocenectomy; Pancreatic fistula; Post-Operative Pancreatic Fistula; Post-Pancreatectomy Acute Pancreatitis; Pancreatic complications; Sepsis; mHLA-DR; Immunparalysis; Immunosuppression
MeSH Terms: conditions — Pancreatic Fistula; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — mHLA-DR analysis will be realized on Cyto-Chex® BCT anticoagulant tubes (5mL). Each sample will be transported and centralized at the Immunology Laboratory of Edouard Herriot Hospital and analyzed by flow cytometry. Results will be expressed as number of receptors per monocyte (Ab/C)
  Samples will be collected :
  * The day of surgery before intervention
  * The day of surgery after intervention
  * At postoperative day one
  * At postoperative day two
  * At postoperative day three
  * At postoperative day four
  * At postoperative day five
  * At postoperative day seven
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults patients undergoing Pancreaticoduodenectomy in one for a benign or malignant tumor of the pan: Biological : blood sample mHLA-DR analysis will be realized on Cyto-Chex® BCT anticoagulant tubes (5mL). Each sample will be transported and centralized at the Immunology Laboratory of Edouard Herriot Hospital and analyzed by flow cytometry. Results will be expressed as number of receptors per monocyte (Ab/C)
  Samples will be collected :
  * The day of surgery before intervention
  * The day of surgery after intervention
  * At postoperative day one
  * At postoperative day two
  * At postoperative day three
  * At postoperative day four
  * At postoperative day five
  * At postoperative day seven
  Interventions: Diagnostic Test: mHLA-DR analysis

INTERVENTIONS:
Diagnostic Test: mHLA-DR analysis — mHLA-DR analysis will be realized on Cyto-Chex® BCT anticoagulant tubes (5mL). Each sample will be transported and centralized at the Immunology Laboratory of Edouard Herriot Hospital and analyzed by flow cytometry.
  Samples will be collected :
  * The day of surgery before intervention
  * The day of surgery after intervention
  * At postoperative day one
  * At postoperative day two
  * At postoperative day three
  * At postoperative day four
  * At postoperative day five
  * At postoperative day seven

SUMMARY:
By 2030, pancreatic adenocarcinoma could become the second leading cause of cancer-related death in France. To date, Pancreaticoduodenectomy (PD) is the standard treatment for resectable adenocarcinoma of the pancreatic head. Despite advances in perioperative care, morbidity remains high, and the occurrence of postoperative complications can negatively impact patient's oncologic prognosis.

Sepsis is the leading cause of postoperative death following PD and it remains mainly associated with the development of a clinically-relevant postoperative pancreatic fistula (CR-POPF). More recently, post-pancreatectomy acute pancreatitis (PPAP) has been defined as a very early complication after pancreatic resection. PPAP is an ischemic and inflammatory condition of the pancreatic remnant that may be responsible for nearly half of CR-POPFs. CR-PPAP can lead to sepsis with multiorgan failure and necrotizing pancreatitis, which are with CR-POPF the two main indications for reoperation and completion pancreatectomy.

Despite the major impact of severe pancreatic complications on mortality after PD, no reliable early biomarker currently exists to predict their occurence.

Immunoparalysis refers to the functional impairment of immune cells with monocytes showing altered capacity of cell presentation. In classical models of inflammation such as acute pancreatitis, sepsis and surgery, the initial systemic inflammatory response syndrome is simultaneously accompanied by a compensatory anti-inflammatory reaction, which may lead to immunoparalysis. mHLA-DR (Human Leukocyte Antigen-DR on Monocytes) is considered as the most appropriate biomarker to assess this immune dysfonction. Various studies emphasize the predictive value of mHLA-DR for early detection of adverse outcomes : in acute pancreatitis, mHLA-DR predicts the onset of severe forms as early as admission and after colorectal surgery, mHLA-DR enables earlier detection of anastomotic leakage compared to conventional biomarkers.

The main hypothesis is that the severity of postoperative complications is driven by immunological factors. On one hand, this study seeks to improve the understanding of the relationship between the immune response after PD and the occurrence of pancreatic complications. On the other hand, it aims to assess if mHLA-DR could represent an early biomarker for detecting severe pancreatic complications.

Therefore, the main objective of this study is to evaluate the association of mHLA-DR expression in the early postoperative period following PD and the occurrence of severe pancreatic complications

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing a Pancreaticoduodenectomy in one of the four participating centers for a benign or malignant tumor of the pancreatic head

Exclusion Criteria:

* Age < 18 years
* Pregnant, postpartum, or breastfeeding women
* Indication other than tumor-related (e.g., chronic pancreatitis)
* Patient with an infectious syndrome at the time of inclusion
* Preoperative immunosuppression
* Immunosuppressive disease other than cancer:

  * Congenital or acquired immune deficiency
  * Functional hyposplenism or asplenia, patient under long-term antibiotic prophylaxis for this reason
  * Patient with HIV (and CD4 < cells/mm³)
  * Aplasia defined by circulating neutrophil count < 500 cells/mm³
  * Immunosuppressive treatment other than chemotherapy : Biotherapy, Corticosteroid therapy >10 mg/day or cumulative dose >700 mg prednisolone equivalent : Patient expected to receive immunosuppressive treatment within the first 7 postoperative days
* Individuals deprived of liberty by judicial or administrative decisio
* Adults under legal protection (guardianship or curatorship)
* Individuals not affiliated with a social security scheme or an equivalent coverage
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients undergoing a Pancreaticoduodenectomy in one of the four participating centers for a benign or malignant tumor of the pancreatic head will be included.
  Participating centers : Hospices Civils de Lyon (Edouard Herriot Hospital, Croix-Rousse Hospital, Lyon Sud Hospital) and Centre Léon Bérard, Lyon, France
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
mHLA-DR expressed by numbers of antibody per cells (Ab/C) | mHLA-DR will be assessed during 7 first days - The day of surgery right before intervention (Pre-Op) - The day of surgery immediately after intervention (Post-Op) - At postoperative day one (POD1) - At postoperative day two (POD2) - At postoperative day
  Association of expression of mHLA-DR at POD1, POD 2 and POD3 and occurrence of pancreatic complications (CR-POPF, CR-PPAP, PACE criteria) PACE (PAncreatic Composite Endpoint) is a binary composite endpoint including : CR-POPF or Hemmorage or Reintervention (endoscopic, radiological, surgical)

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Julie PERINEL, Lyon
  - Xavier MULLER, Lyon
  - Aurélien DUPRE, Lyon
  - Jean-Christophe LIFANTE, Pierre-Bénite